#### **Informed consent form**

Document date: January 1, 2024

#### Research title

Clean Catch Urine Feasibility and Contamination Rate compared to Bladder Catheterization Urine in Pre-Continent Children: Randomized Control Trial

### Research Idea

Our study aims to test an alternative way to urine collection by catheterization. primary outcomes are to compare the contamination rates between the two method and parent satisfaction. The secondary outcomes, include procedure duration, pain score (using neonatal infant pain scale)

# Methodology

The patient will be randomly distributed into two groups: group one, urine will be collected through catheterization, group two urine will be collected by Clean Catch urine collection.

## **Contact information**

If you have any questions, you may ask now or later, even after the study has started. If you wish to ask questions later, you may contact any of the following: -Dr.Sulayyem Al Hasrousi, contact number +968 97383155, E-Mail: alharsoosi@gmail.com.

- Dr. Dr. Muna Al Ka'abi, contact number +968 91797366, E-Mail: r2126@resident.omsb.org
- I am the parent of .....
- I have read the foregoing information, or it has been read to me. I have had the opportunity to ask questions about it.
- Any questions that I asked, they have been answered to my satisfaction. I consent voluntarily to participate as a participant in this research.

Authorized to consent name: Relationship to the patient: Signature date:

Researcher/Doctor: